CLINICAL TRIAL: NCT04645654
Title: A Randomized-controlled Clinical Trial of Brief Postoperative Hypnosis Intervention as Multimodal Analgesia After Major Abdominal Surgery in the ERAS Protocol
Brief Title: Brief Postoperative Hypnosis Intervention as Multimodal Analgesia After Major Abdominal Surgery
Acronym: Hypn+ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Chantal Berna, Professor, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-VD 2020-01710
Record Dates: First submitted 2020-11-13; First posted 2020-11-27 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Hypnosis; ERAS; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis (Experimental): 3 sessions of script-based hypnosis (analgesic suggestions) + recordings provided for self-hypnosis
  Interventions: Behavioral: Hypnosis
- Standard of care (No Intervention): Standard of care ERAS based optimized multimodal analgesia, without any complementary medicine

INTERVENTIONS:
Behavioral: Hypnosis — Three sessions of 30 minute hypnosis, based on standardised script, focused on pain management.
  Arms: Hypnosis

SUMMARY:
This study will measure the efficacy of hypnosis on pain after a major abdominal surgery. The aim is to further improve comfort and rehabilitation of patients after surgery, beyond the usual early recovery after surgery (ERAS) enhancement protocols.

Patients will be randomised (1:2) to the standard of care regarding pain management and rehabilitation, as part of the ERAS protocol, vs. ERAS + an additional hypnosis intervention. In this group, hospitalised patients are given 3 hypnosis sessions targeting analgesia between postoperative day 1 to 12.

The study will collect outcomes about pain and its burden, sleep quality, appetite, mobilisation and mood. Secondary outcomes also include use of pain medication and length of hospital stay.

DETAILED DESCRIPTION:
The primary objective of the present study is to evaluate the efficacy of hypnosis as an adjunct to the standard of care pain management program on postoperative pain compared to the standard ERAS program. Our hypothesis is that hypnosis, as part of a multi-modal analgesic management plan, will lead to decreased levels of pain compared to standard of care.

A secondary hypothesis is that better controlled pain will lead to enhanced recovery, in terms of post-operative incidence of complications, physical comfort and independence, psychological and emotional state and length of stay.

This study is an open label randomized controlled trial with two arms, comparing hypnosis as adjunctive therapy vs. standard of care. It is a monocentric study and will take place at Centre Hospitalier Universitaire Vaudois (CHUV), a teaching hospital in Lausanne, Switzerland. It represents a collaboration between the Service of Visceral Surgery and the Center of Integrative and Complementary Medicine.

Participants will be recruited before a planned surgery, as well as in the post-surgical setting. They will be screened by the study team to ensure they fulfil the inclusion criteria. If eligible and after informed consent is obtained, an assessment of the cognitive function will be performed (cf. Chapter 4: study population). All included participants will then be randomized in a 2:1 proportion to the "Hypnosis (H)" group or the "Standard of Care (SOC)" group.

After major abdominal surgery, all participants will benefit from a standard ERAS recovery program. The ERAS protocol involves multimodal pain management with medications, interventional pain therapy as needed, and psychological support if needed.

Relevance:

Acute pain has a major impact on LOS after surgery due to delayed recovery and opioid side effects. Furthermore, acute pain represents a risk for chronic pain, with its massive impact on quality of life and function. Interest is growing for non-pharmacological interventions as part of a multimodal approach for acute pain management. Hypnosis could be a low risk, cost-effective complementary therapy to improve patients' pain management, with possible impact on recovery and eventually a reduction of the length of hospital stay after surgery. If hypnosis is demonstrated to be an effective way to improve post-operative pain management in fragile patients undergoing massive abdominal surgery, then this therapy could be offered more broadly as adjunction to the actual standard of care in our teaching hospital.

Furthermore, the Department of Visceral Surgery at CHUV is a teaching ward, accredited by the ERAS society. Therefore, results may be used to improve patient care within the ERAS society more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adults (from 18 years old).
* Major abdominal surgery with planned hospitalisation of more than seven days post-operatively, according to clinician's evaluation
* Able to give informed consent as documented by signature
* Interested in trying hypnosis as a complementary pain management therapy

Exclusion Criteria:

* Inability to engage in the intervention of the study, e.g. inability to communicate in French without a translator, cognitive impairment, severe hearing impairment
* Acute psychiatric (e.g. psychotic or suicidal ideation) or somatic (e.g. unstable cardio-respiratory condition) co-morbidity preventing full engagement during intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity at mobilisation | Between postoperative day 1 to 12.
  visual analogue pain intensity scale from 0 (no pain) to 10 (most intense pain imaginable)

SECONDARY OUTCOMES:
Pain intensity at rest | Between postoperative day 1 to 12.
  visual analogue pain scale from 0 (no pain) to 10 (most intense pain imaginable)
Pain unpleasantness | Between postoperative day 1 to 12.
  visual analogue scale from 0 (not unpleasant) to 10 (most unpleasant pain imaginable)
Opioid consumption | Between postoperative day 1 to 12
  opioid name and dose (mg) recorded in medical chart
Post-surgical complications | Between postoperative day 1 to 12
  list of complications recorded in patient's medical chart
Length of hospital stay | through study completion; records checked up to 100 days after end of study participation
  date of entry to date of release from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Berna, Prof, Principal Investigator — Centre de médecine intégrative et complémentaire, CHUV
Locations (1):
- Centre de Médecine Intégrative et Complémentaire, CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No